CLINICAL TRIAL: NCT01047605
Title: Evaluation of the Pharmacological Effects of NEURAPAS® Balance and PASCOFLAIR® 425 mg by Quantitative Measurement of Brain Activity in 16 Healthy Volunteers. A Single-blinded, Randomised, Placebo-controlled, 3-armed Phase-I-study With Cross-over Design
Brief Title: Pharmacological Effects of Neurapas® Balance and Pascoflair® 425 mg on Brain Activity in Healthy Volunteers
Acronym: NCAG 5209
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Responsible Party: Anja Braschoss, MD, PASCOE pharmazeutische Praeparate GmbH
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 173 S 09 PSY; 2009-015827-97 (EudraCT Number)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Healthy
Keywords: qEEG; herbal medicine; cognitive function; Neurapas balance; Pascoflair; hypericum; passionflower; valerian; Healthy volunteers; Influence on quantitative electro-encephalogram (qEEG).

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- PP1 (Experimental): Neurapas balance
  Interventions: Drug: Neurapas balance
- PP2 (Experimental): Pascoflair 425 mg
  Interventions: Drug: Pascoflair 425 mg
- PL1 (Placebo Comparator): P-Tabletten weiß
  Interventions: Drug: P-Tabletten weiß

INTERVENTIONS:
Drug: Neurapas balance — 6 tablets single dose
  Arms: PP1
Drug: Pascoflair 425 mg — 3 tablets , single dose
  Arms: PP2
Drug: P-Tabletten weiß — 3 tablets, single dose
  Arms: PL1

SUMMARY:
To evaluate the pharmacological effects of two herbal medicinal products (Neurapas balance and Pascoflair 425 mg) in comparison to placebo on brain activity.

DETAILED DESCRIPTION:
Evaluation of the pharmacological effects of Neurapas® balance and Pascoflair® 425 mg by quantitative measurement of brain activity in 16 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers
* 30 - 70 years (extremes included)
* Medical history without any study relevant pathological findings
* Written and signed informed consent

Exclusion Criteria:

* Clinically study relevant acute or chronic disorders, that can be detected by clinical investigation or medical history
* Clinical, study-relevant pathological findings of clinical oar laboratory investigations
* Clinically relevant pathological EEG findings (e.g. artefact-free parts in Screening-EEG <30% in one recording
* Clinically relevant allergies
* positive alcohol testing on Screening, Day A, B, or C, or anamnestic
* positive drug screening test on Screening, Day A, B, or C, or anamnestic
* Intake of study relevant medication 14 days prior to active Day A, or during active study duration, based on the volunteer´s information
* Regular intake of drug with primary central nervous effects (e.g. psychoactive drugs or central acting antihypertensive drugs)
* Known hypersensitivity / allergy against herbal extracts (i.e. dry extracts of Passionflower herb, St. John´s Wort herb, Valerian root) or lactose or an other excipient of the investigational medication
* Lapp-lactase deficiency (anamnestic)
* Hypersensitivity of the skin (anamnestic)
* BMI (Body-Mass-Index) <18 or>30
* Abuse of caffeine, teeine, or tobacco
* Smoking in the investigational site on Day A, B, or C
* Participation in an other clinical study within 60 days prior to Screening
* Positive Pregnancy Test (on Screening, Day A, B, or C) or Lactation
* Bad compliance
* Revocation of informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Z1: qEEG (total): Median change of electrical activity (qEEG: of all electrode positions) compared to Baseline (PP1 vs PP2 vs Placebo) | 5 times within 4 h

SECONDARY OUTCOMES:
Comparison PP1 vs PP2 vs Placebo: Z2: qEEG (all frequencies, Clusters): Median change of electrical activity (qEEG: of selective brain-regional clusters of electrode positions) compared to Baseline | 5 times within 4 h
Comparison PP1 vs PP2 vs Placebo: Z3:qEEG (d2, beta1 (Cluster F7/T3)) | 5 times wihtin 4 h
Comparison PP1 vs PP2 vs Placebo: Z4:qEEG (ME, theta (Cluster F7/T3/T6)) | 5 times within 4 h
Comparison PP1 vs PP2 vs Placebo: Z5:qEEG (KLT, theta (Cluster F7/T3) + alpha (Cluster T4/T6)) | 5 times within 4 h
Comparison PP1 vs PP2 vs Placebo: Z6: qEEG (Aa, all frequencies, Cluster C3/T3/P4) | 5 times within 4 h
Comparison PP1 vs PP2 vs Placebo: Z7: Timely onset of effect and duration of effect | 5 times within 4 h

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Wedekind, MD, PhD, Principal Investigator — Neurocoed AG, Sportparkstr. 9, D-35578 Wetzlar, Germany; Wilfried Dimpfel, Prof, Study Chair — Neurocode AG, Sportparkstr. 9, D-35578 Wetzlar, Germany; Anja Braschoss, MD, Study Director — Pascoe Pharmazeutische Praeparate GmbH
Locations (1):
- Neurocode AG, Wetzlar, Germany

REFERENCES:
- [Derived] Dimpfel W, Koch K, Weiss G. Early effect of NEURAPAS(R) balance on current source density (CSD) of human EEG. BMC Psychiatry. 2011 Aug 2;11:123. doi: 10.1186/1471-244X-11-123. PMID 21810233